CLINICAL TRIAL: NCT01750879
Title: Clinical Desensitization and Tolerance Following Peanut Oral Immunotherapy and Subsequent Allergen Avoidance
Brief Title: Tolerance Following Peanut Oral Immunotherapy
Acronym: PNOIT2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Wayne G. Shreffler, MD, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2012P002153; 5U19AI095261-02 (NIH)
Record Dates: First submitted 2012-12-13; First posted 2012-12-17 (Estimated); Results first posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Peanut Allergy
Keywords: peanut; allergy; food; immunotherapy; tolerance; desensitization
MeSH Terms: conditions — Peanut Hypersensitivity; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peanut Flour (Active Comparator): Oral Immunotherapy with peanut flour.
  Interventions: Drug: Peanut Flour
- Oat Flour (Placebo Comparator): Oral Immunotherapy with oat flour.
  Interventions: Drug: Oat Flour

INTERVENTIONS:
Drug: Peanut Flour — Peanut Flour
  Arms: Peanut Flour
Drug: Oat Flour — Oat Flour
  Arms: Oat Flour

SUMMARY:
The unifying objective of this project is to determine whether peanut oral immunotherapy (PN OIT) induced clinical tolerance in the context of food allergy is significantly associated with the expansion of a specific regulatory T cell subset (CD45RA- CD25++ FoxP3++) that is thought to be inducible in the gut-associated lymphoid compartment and associated with immunological tolerance.

The hypothesis of the study is that the induction of Treg cells will be associated with clinical tolerance.

The investigators will measure the change from baseline of induced Treg cells as a frequency of total CD4 T cells during active treatment and compare that between participants who achieve significant clinical tolerance (Tolerance and Partial Tolerance Groups as defined below) and those who do not (Treatment Failure Group).

DETAILED DESCRIPTION:
Clinical Objectives:

1. To evaluate whether PN OIT induces increased tolerance, defined as a statistically significant increase in the median eliciting dose (ED) from a double-blind placebo-controlled food challenge (DBPCFC) before and after treatment with PN OIT and after subsequent allergen avoidance.
2. To evaluate whether PN OIT induces clinical desensitization, defined as 1) a median 10-fold or greater increase in ED at DBPCFC before and after PN OIT treatment period 2) a statistically significant higher median ED at DBPCFC following treatment period between active and control treatment; and 3) a significantly lower frequency of accidental ingestion reactions in active versus control treatment.
3. To evaluate the safety of PN OIT.

Mechanistic Objectives:

1. To determine whether PN OIT induces a statistically significant increase in the TCR clonal diversity of Treg populations during active treatment among participants who achieve increased clinical tolerance (Tolerance and Partial Tolerance Groups as defined in clinical endpoints) versus the Treatment Failure Group.
2. To determine whether PN OIT suppresses mast cells by inducing a significant suppression of the median ED on end-point dilution skin testing in actively treated participants by the end of maintenance therapy.
3. To determine whether PN OIT suppresses basophils as defined by a 10-fold suppression of peanut-specific basophil ED in actively treated participants by end of a maintenance period.
4. To determine whether either mast cell or basophil suppression at the end of maintenance therapy is significantly associated with clinical outcomes following avoidance.

Exploratory Objectives:

1. To describe the gene expression profiles and clonal diversity of regulatory and effector T cell subsets before and after OIT to better understand the phenotype and ontogeny of these subsets and potentially discover new therapeutic pathways.
2. To engineer human MHC class II tetramers on common HLA backgrounds and map T cell epitopes of the dominant peanut allergens for use in validating earlier findings and for future studies of peanut-specific immune responses in humans.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of peanut allergy by a positive skin prick test to peanut (reaction wheal at least 5 mm larger than saline control) and by medical history or Serum peanut-specific IgE >5 kU/L at screening visit.
* Ara h 2 specific IgE >0.35 kU/L at screening visit
* Ability to provide informed consent.
* Males and females of all ethnic/racial groups aged 7-55 years old who are otherwise healthy.
* React to less than 443 mg of peanut protein during DBPCFC1

Exclusion Criteria:

* History of severe anaphylaxis as defined by hypoxia (cyanosis or SpO2 <92% during reaction), documented hypotension (documented systolic BP >30% below predicted normal for sex, height, weight or from known baseline), neurological compromise (confusion, loss of consciousness), or incontinence.
* Severe or Moderate asthma as defined using the severity criteria of the current NHBLI Guidelines for the Diagnosis and Management of Asthma (http://www.nhlbi.nih.gov/guidelines/asthma/).
* Poorly-controlled asthma as defined by FEV1 <80% or any of the following symptoms: nighttime awakening >2 days/week or rescue medication use >2 days / week.
* Diagnosis of other severe or complicating medical problems, including autoimmune or chronic immune inflammatory conditions or gastrointestinal inflammatory conditions, including Celiac Disease, Inflammatory Bowel Disease and Eosinophilic Gastrointestinal Disorders
* Inability to cooperate with and/or perform oral food challenge procedures.
* Primary Immune Deficiency
* Allergy to oat confirmed by skin prick testing and history
* Current use of beta blockers, angiotensin converting enzyme inhibitors, or monoamine oxidase inhibitors
* Women of childbearing potential who are pregnant, planning to become pregnant, or breastfeeding
* Hemoglobin level less than 12.5 gm/dL at screening. Weight <23 kg
* Use within the past 6 months of other systemic immunomodulatory treatments including allergen immunotherapy, or use of biologics with an immune target, including omalizumab.
* Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study may also exclude a participant from the study.

Ages: 7 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2013-08; Primary Completion 2017-07-11 (Actual); Study Completion 2017-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wayne G Shreffler, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
de-identified data exported from REDCap
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: upon request within the year and without planned time limitation

REFERENCES:
- [Derived] Monian B, Tu AA, Ruiter B, Morgan DM, Petrossian PM, Smith NP, Gierahn TM, Ginder JH, Shreffler WG, Love JC. Peanut oral immunotherapy differentially suppresses clonally distinct subsets of T helper cells. J Clin Invest. 2022 Jan 18;132(2):e150634. doi: 10.1172/JCI150634. PMID 34813505

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from a specialty clinic, college campus clinic, and community outreach (including advertisements on Boston MBTA) between May 2013 and January 2016. The first participant was enrolled in August 2013.
Pre-assignment Details: 113 screened, 72 excluded (3 Lost to follow-up pre-randomization; 8 Re-screened following protocol change; 21 Screen Fail no objective symptoms on DBPCF1; 29 Screen Fail prior to DBPCFC; and 11 Voluntary withdrawal pre-randomization)
Groups:
- Peanut Flour: Participants will be randomly assigned by study statistician to treatment or placebo groups at a ratio of 3:1 following a double-blind placebo controlled food challenge, DBPCFC1, on 2 separate days. One challenge will consist of 5 doses of peanut in increasing amounts up to a total of 443 mg of peanut protein masked in vehicle food. The second day will consist of placebo material given similarly. Participants with an eliciting dose of 443mg or less will receive daily escalating dosages of peanut flour OIT in a blinded fashion, as described in the modified rush phase, until a daily dose of 4000 mg is reached. Following treatment, a 2nd challenge will occur DBPCFC2, identical to DBPCFC1, but with additional doses of 1000 mg and 3000 mg for a cumulative dose of 4443 mg peanut protein. After 12 weeks of complete peanut avoidance, participants will undergo a third challenge, DBPCFC3, which will follow a slightly different schedule of doses for a cumulative dose of 4430 mg peanut protein.
- Placebo (Oat) Flour: Participants in the placebo arm will follow the same protocol except they receive daily escalating dosages of placebo oat flour, and they will not participate in DBPCFC3. Following DBPCFC2, assignment will be unblinded and placebo participants will be offered open-label active treatment under a separate protocol.
Period: Overall Study
Arm/Group | Peanut Flour | Placebo (Oat) Flour
Started | 30 | 11
DBPCFC2 | 20 | 8
DBPCFC3 | 20 | 0
Completed | 20 | 8
Not Completed | 10 | 3
Not completed — Adverse Event | 8 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Did not complete per protocol | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Active: Participants will be randomly assigned by study statistician to treatment or placebo groups at a ratio of 3:1 following a double-blind placebo controlled food challenge, DBPCFC1, on 2 separate days. One challenge will consist of 5 doses of peanut in increasing amounts up to a total of 443 mg of peanut protein masked in vehicle food. The second day will consist of placebo material given similarly. Participants with an eliciting dose of 443mg or less will receive daily escalating dosages of peanut flour OIT in a blinded fashion, as described in the modified rush phase, until a daily dose of 4000 mg is reached. Following treatment, a 2nd challenge will occur DBPCFC2, identical to DBPCFC1, but with additional doses of 1000 mg and 3000 mg for a cumulative dose of 4443 mg peanut protein. After 12 weeks of complete peanut avoidance, participants will undergo a third challenge, DBPCFC3, which will follow a slightly different schedule of doses for a cumulative dose of 4430 mg peanut protein.
- Placebo: Participants in the placebo arm will follow the same protocol except they receive daily escalating dosages of placebo oat flour, and they will not participate in DBPCFC3. Following DBPCFC2, assignment will be unblinded and placebo participants will be offered open-label active treatment under a separate protocol.
- Total: Total of all reporting groups
Arm/Group | Active | Placebo | Total
Number analyzed (Participants) | 30 | 11 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 7 | 21
  Between 18 and 65 years | 16 | 4 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 20.5 (11.1) | 16.3 (7.2) | 19.4 (10.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 18 | 5 | 23
  Male | 11 | 6 | 17
  Transgender | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 27 | 11 | 38
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 24 | 10 | 34
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 30 | 11 | 41
Peanut-specific IgE [Mean (Standard Deviation); unit: kU/L] | 116 (156) | 97.5 (121) | 111.3 (146.4)

OUTCOME MEASURES:

1. Primary Outcome: Tolerance, Partial Tolerance, or Treatment Failure
Description: 1. Tolerance: Ingestion of 4430 mg of peanut protein at DBPCFC3 without symptoms.
  2. Partial Tolerance: ED at DBPCFC3 <4430 mg but =>430 mg AND >10-fold more than at DBPCFC1.
  3. Treatment Failure - non desensitized: Failure to achieve the minimum maintenance dose (600 mg) of peanut protein by 12 months, or an ED <1443 mg at DBPCFC2, or ED at DBPCFC3 <443 mg OR <10-fold more than at DBPCFC1.
  4. Treatment Failure - withdrawal
Time Frame: Average 515 days from DBPCFC1 to DBPCFC3
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Placebo
Number analyzed (Participants) | 30 | 11
Participants
  Tolerance | 5 | 0
  Partial Tolerance | 8 | 0
  Treatment Failure- non-desensitized | 7 | 8
  Treatment Failure- withdrawal | 10 | 3

2. Secondary Outcome: Clinical: Tolerance
Description: The change in median eliciting dose (ED) from DBPCFC1 to DBPCFC3. (note: ED right censored to maximum dose for those without any clinical reactivity)
Time Frame: 630 days
Population: Per protocol, subjects were unblinded after DBPCFC2 and those on placebo were not subjected to DBPCFC3
Measure: Median (Full Range); unit: mg
Arm/Group | Peanut Flour | Placebo (Oat) Flour
Number analyzed (Participants) | 20 | 0
mg | 4000 [-403 to 4400] |

3. Secondary Outcome: Clinical: Desensitization
Description: - The change in median eliciting dose (ED) from DBPCFC1 to DBPCFC2.
Time Frame: 518 days
Population: 30 active and 11 placebo had baseline challenge (DBPCFC1); 20 active and 8 placebo had first post-treatment challenge (DBPCFC2). Change in median eliciting dose restricted to the 20 and 8 who competed DBPCFC2 (i.e., per protocol)
Measure: Median (Full Range); unit: mg
Arm/Group | Peanut Flour | Placebo (Oat) Flour
Number analyzed (Participants) | 20 | 8
mg | 4000 [-3 to 4400] | -65 [-430 to 500]

4. Secondary Outcome: Clinical: Safety
Description: - The rate of reported adverse advents due to accidental ingestions in the active versus placebo groups.
Time Frame: 630 days
Measure: Count of Participants; unit: Participants
Arm/Group | Peanut Flour | Placebo (Oat) Flour
Number analyzed (Participants) | 30 | 11
Participants | 0 | 0

5. Secondary Outcome: Mechanistic: TCR Clonal Diversity
Description: The change in the TCR clonal diversity of in vitro allergen-expanded Treg cells and induced Treg cells measured by TCRB CDR3 sequence clonotyping of sorted cells during active treatment among participants who achieve increased clinical tolerance (Tolerance and Partial Tolerance Groups as defined in clinical endpoints) versus the Treatment Failure Group.
  We conducted a nested case-control analysis of a subset of actively treated (by treatment outcome) versus placebo treated patients. Genomic DNA was used to amplify and sequence the complementarity-determining region 3 (CDR3) regions (immunoSEQ assay; Adaptive Biotechnologies).
  Enriched clonotypes in the CD154+ fraction (doi: https://doi.org/10.1101/2020.05.11.088286) were analyzed for differences by Rank Abundance Curve analysis (R package alakazam; Chao A, et al. Ecology. 2015 96, 11891201) to determine differences in clonal diversity.
Time Frame: 630 days
Population: We conducted a nested case-control analysis of a subset of actively treated (by treatment outcome) versus placebo treated patients. Genomic DNA was used to amplify and sequence the complementarity-determining region 3 (CDR3) regions (immunoSEQ assay; Adaptive Biotechnologies). Enriched clonotypes in the CD154+ fraction (doi: https://doi.org/10.1101/2020.05.11.088286) were analyzed for differences by Rank Abundance Curve analysis (R package alakazam; Chao A, et al. Ecology. 2015 96, 11891201).
Measure: Mean (95% Confidence Interval); unit: percentage of clones
Groups:
- Peanut Flour -- Tolerance: Tolerance: Ingestion of 4430 mg of peanut protein at DBPCFC3 without symptoms.
- Peanut Flour -- Partial Tolerance: Partial Tolerance: ED at DBPCFC3 <4430 mg but ≥430 mg AND >10-fold more than at DBPCFC1.
- Peanut Flour -- Treatment Failure: Treatment Failure: Inability to tolerate the minimum maintenance dose (600 mg) of peanut protein by 12 months, or an ED <1443 mg at DBPCFC2, or ED at DBPCFC3 <443 mg OR <10-fold more than at DBPCFC1
- Placebo: Placebo (Oat Flour) treated participants.
Arm/Group | Peanut Flour -- Tolerance | Peanut Flour -- Partial Tolerance | Peanut Flour -- Treatment Failure | Placebo
Number analyzed (Participants) | 5 | 6 | 6 | 5
percentage of clones | 0.010499258 [0.0061792665 to 0.014819249] | 0.003841910 [0.0011267402 to 0.006557080] | 0.003090797 [0.0007072315 to 0.005474362] | 0.003592776 [0.0009671402 to 0.006218412]

6. Secondary Outcome: Mechanistic: Change Eliciting Dose of End-point Dilution.
Description: The change in eliciting dose of end-point dilution skin testing between actively treated and placebo treated participants following maintenance therapy and the change in ED of end-point dilution skin testing among actively treated participants following maintenance therapy and avoidance between clinical outcome groups.
Time Frame: 518 days
Population: skin test quality was poor
Arm/Group | Peanut Flour | Placebo (Oat) Flour
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Mechanistic: Change in Basophil Eliciting Dose.
Description: The change in peanut-specific basophil ED in actively treated participants at the end of maintenance and the end of avoidance between clinical outcome groups.
Time Frame: 630 days
Population: basophil time points inadequate for analysis
Arm/Group | Peanut Flour | Placebo (Oat) Flour
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Mechanistic: Change in Peanut Allergen-specific IgG4
Description: The change in peanut allergen-specific IgG4 in actively treated participants by the end of maintenance between clinical outcome groups.
Time Frame: 518 days
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Peanut Flour | Placebo (Oat) Flour
Number analyzed (Participants) | 22 | 9
mg/mL | 0.664 (0.559) | 0.375 (0.247)

9. Secondary Outcome: Mechanistic: Significant Gene Expression Changes by Transcriptional Profiling of Regulatory and Effector T Cell Populations
Description: Statistically significant gene expression changes (as number of genes) by transcriptional profiling of regulatory and effector T cell populations before and after OIT between clinical outcome groups.
  Total RNA from CD154+ and CD154-CD69- T cells was used for cDNA synthesis and amplification. Libraries were prepared and sequenced to a read depth of approximately 30 million reads per sample (Illumina HiSeq) and aligned to the hg19 human reference genome with the ensemble version 75 annotation using STAR version 2.5.3a,(Dobin et al. Bioinformatics 2013) and gene expression was summarized using RSEM version 1.3.0 (Li et al. BMC Bioinform 2013). Differential expression analysis was performed using DESeq2 v 1.30.1 (R v 4.04). Significance level was set at an unadjusted P value less than .001.
Time Frame: 630 days
Population: Subjects as defined per protocol. All 5 placebo were 'treatment failure -- non-desensitized' and per protocol, none were eligible for avoidance or DBPCFC3.
  Total RNA from CD154+ and CD154-CD69- T cells was used for cDNA synthesis and amplification. Read depth of approximately 30 million per sample (Illumina HiSeq) and aligned to the hg19 human reference genome with the ensemble version 75 annotation. Differential expression analysis was performed using DESeq2 v 1.30.1 (R v 4.04).
Measure: Number; unit: number of differentially expressed genes
Groups:
- Peanut Flour - Tolerance: Tolerance: Ingestion of 4430 mg of peanut protein at DBPCFC3 without symptoms.
- Peanut Flour - Treatment Failure: Treatment Failure: Inability to tolerate the minimum maintenance dose (600 mg) of peanut protein by 12 months, or an ED <1443 mg at DBPCFC2, or ED at DBPCFC3 <443 mg OR <10-fold more than at DBPCFC1.
- Peanut Flour - Partial Tolerance: Partial Tolerance: ED at DBPCFC3 <4430 mg but ≥430 mg AND >10-fold more than at DBPCFC1.
- Placebo - Treatment Failure: Received oat flour (placebo) treatment. All treatment failures; 3 due to early withdraw, 8 by DBPCFC2 outcome. Per protocol, none advanced to DBPCFC3.
Arm/Group | Peanut Flour - Tolerance | Peanut Flour - Treatment Failure | Peanut Flour - Partial Tolerance | Placebo - Treatment Failure
Number analyzed (Participants) | 5 | 6 | 6 | 5
number of differentially expressed genes
  genes up at maintenance versus baseline | 86 | 45 | 12 | 9
  genes up at avoidance versus baseline | 42 | 14 | 43 | NA — not evaluable per protocol
  genes down at maintenance versus baseline | 43 | 154 | 18 | 3
  genes down at avoidance versus baseline | 9 | 39 | 15 | NA — not evaluable per protocol

ADVERSE EVENTS:
Time Frame: August 2013 to January 2016 (2 years and 5 months)
Description: Build up AEs, At home AEs, DBPCFC2 AEs
Arm/Group | Peanut Flour | Oat Flour
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/11
Other Adverse Events (participants affected / at risk) | 30/30 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peanut Flour (N=30) | Oat Flour (N=11)
Suicidal Ideation, unrelated (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Peanut Flour (N=30) | Oat Flour (N=11)
Anaphylactic Reaction (Immune system disorders) | 5 (12) | 1 (1) — Build up AEs; Moderate to severe AEs reported
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) — Build up AEs; Moderate to severe AEs reported
Nausea/Vomting (Gastrointestinal disorders) | 1 (1) | 0 (0) — Build up AEs; Moderate to severe AEs reported
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) — At home AEs; Moderate to severe AEs reported
Anaphylactic Reaction (Immune system disorders) | 15 (89) | 0 (0) — At home AEs; Moderate to severe AEs reported
Abdominal Pain (Gastrointestinal disorders) | 4 (17) | 0 (0) — At home AEs; Moderate to severe AEs reported
Nausea/Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) — At home AEs; Moderate to severe AEs reported
Asthma Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) — At home AEs; Moderate to severe AEs reported
Skin/oral pruritis (Immune system disorders) | 1/20 (1) | 2/9 (2) — DBPCFC2 AEs; 20 subjects on peanut; 9 subjects on placebo
Angiodema (Skin and subcutaneous tissue disorders) | 1/20 (1) | 0/9 (0) — DBPCFC2 AEs; 20 subjects on peanut; 9 subjects on placebo
Anaphylactic Reaction (Immune system disorders) | 7/20 (7) | 7/9 (7) — DBPCFC2 AEs; 20 subjects on peanut; 9 subjects on placebo
Reflux (Gastrointestinal disorders) | 1/20 (1) | 0/9 (0) — DBPCFC2 AEs; 20 subjects on peanut; 9 subjects on placebo
Abdominal Pain (Gastrointestinal disorders) | 1/20 (1) | 1/9 (1) — DBPCFC2 AEs; 20 subjects on peanut; 9 subjects on placebo
Nausea/Vomiting (Gastrointestinal disorders) | 0/20 (0) | 1/9 (1) — DBPCFC2 AEs; 20 subjects on peanut; 9 subjects on placebo
Other (Gastrointestinal disorders) | 0/20 (0) | 1/9 (1) — DBPCFC2 AEs; 20 subjects on peanut; 9 subjects on placebo
Wheeze/SOB (Respiratory, thoracic and mediastinal disorders) | 0/20 (0) | 1/9 (1) — DBPCFC2 AEs; 20 subjects on peanut; 9 subjects on placebo

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-29): https://cdn.clinicaltrials.gov/large-docs/79/NCT01750879/Prot_SAP_000.pdf